CLINICAL TRIAL: NCT06262152
Title: Characterization of Sleep Features in Pediatric Patients With Septa-optic Dysplasia
Brief Title: Sleep Profile of Patients With Septo-optic Dysplasia
Status: Recruiting | Type: Observational
Sponsor: IRCCS National Neurological Institute "C. Mondino" Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 49187/2023
Record Dates: First submitted 2024-01-30; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Septo-Optic Dysplasia; Agenesis of Corpus Callosum; Blindness
Keywords: sleep; actigraphy; brain malformation; visual deficit; SOD; genesis of corpus callous; pediatric patients
MeSH Terms: conditions — Septo-Optic Dysplasia; Agenesis of Corpus Callosum; Blindness; Vision Disorders | interventions — Actigraphy; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood; saliva
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Septo-optic dysplasia, visual deficit and agenesis of corpus callosum: * age 3-18 years
  * availability of at least 2 serial sleep EEGs performed during clinical follow-up
  * stable drug therapy in the last three months
  Interventions: Diagnostic Test: Actigraphy, blood and salivary sample, and sleep evaluation

INTERVENTIONS:
Diagnostic Test: Actigraphy, blood and salivary sample, and sleep evaluation — * For each subject, one 4 mL blood and one 2 mL saliva samples will be collected at each assessment.
  * 7 days actigraph recording through wearing of Actiwatch spectrum plus at home
  * Standardized sleep questionnaire administration

SUMMARY:
The aim of this study is to evaluate sleep of patients with septo-optic dysplasia compared to patients with an isolated disorder of peripheral visual system and patients with corpus callosum agenesis since both visus defict and agenesis of corpus callosum might be present SOD but associated to other features / structural and functional anomalies.

Included patients and their caregivers will be asked to compile standardize sleep questionnaires and a sleep screening through an interview will be scheduled. Patients will be asked to wear an actigraph on their non-dominant hand wrist for 7 days.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate sleep of patients with septo-optic dysplasia compared to patients with an isolated disorder of peripheral visual system and patients with corpus callosum agenesis since both visus defict and agenesis of corpus callosum might be present SOD but associated to other features / structural and functional anomalies.

The secondary aims of this study are the following:

1. identify which factors such as clinical and neuroanatomical features including sensory experience influence sleep outcome and how
2. describe melatonin profile of patients with SOD
3. describe sleep EEG of patients with SOD

Three groups of patients will be included:

* Group A: patients with septo-optic dysplasia
* Group B: patients with disorder of peripheral visual system
* Group C: patients with Corpus Callosum agenesis

This is an observational monocentric study. The procedures in the study that are not included in current clinical practice in the follow-up pathway of the included patients are the following:

* administration of standardized sleep questionnaires (Pittsburgh Sleep Quality Index: self-completed questionnaire assessing sleep quality over a 1-month time interval;Epworth Sleepiness Scale: self-completed questionnaire assessing daytime sleepiness; Children sleep habits questionnaire)
* 7 days actigraph recording through wearing of Actiwatch spectrum plus at home
* Performance of Sleep EEG
* Performance of blood and salivary sampling for melatonin dosing (for each subject, one 4 mL blood and one 2 mL saliva samples will be collected at each assessment)

ELIGIBILITY:
Inclusion criteria group A:

* diagnosis of SOD or SOD plus syndrome with or without a defined genetic diagnosis
* age 3-18 years
* availability of at least 2 serial sleep EEGs performed during clinical follow-up
* stable drug therapy in the last three months

Inclusion criteria group B:

* diagnosis of congenital or early acquired isolated peripheral visual deficit with or without a known genetic diagnosis (e.g., congenital cataract, inherited retinal dystrophies, isolated eye maldevelopment).
* age 3-18 years
* grating or visual acuity < 3/10
* availability of serial sleep EEGs performed during clinical follow-up
* stable drug therapy in the last three months

Inclusion criteria group C

* isolated corpus callosum agenesis at brain MRI
* age 3-18 years
* availability of at least 2 serial sleep EEGs performed during clinical follow-up
* stable drug therapy in the last three months

Exclusion criteria group A:

* absence of informed consent
* severe Intellectual disability and/or severe motor impairment
* melatonin assumption

Exclusion criteria group B:

* absence of informed consent
* CNS involvement ( malformations/ lesions)
* severe Intellectual disability and/or severe motor impairment
* melatonin assumption

Exclusion criteria group C

* absence of informed consent
* severe Intellectual disability and/or severe motor impairment
* melatonin assumption

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Three groups of patients will be included:
  * Group A: 15 patients with septo-optic dysplasia
  * Group B: 15 patients with disorder of peripheral visual system
  * Group C: 15 patients with Corpus Callosum agenesis
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2025-05-20 (Estimated)

PRIMARY OUTCOMES:
Sleep profile ( Sleep quality, sleep efficiency) of patients with SOD | 12 months
  SLEEP QUALITY will be assessed through standardized questionnaires :Pittsburgh Sleep Quality Index: self-completed questionnaire ;Epworth Sleepiness Scale: self-completed questionnaire assessing daytime sleepiness; Children sleep habits questionnaire .
  Sleep quality and sleep-wake cycle will be evaluated, namely Child's inability to go to bed, the delay in falling asleep, sleep duration, overnight awakenings, anxiety related to sleep, parasomnia, respiratory disorders, and daytime sleepiness.
  SLEEP EFFICIENCY will be measured by actigraphic assessment of sleep efficiency (the ratio of total sleep time to sleep period), total nighttime sleep duration, rest activity and number of awakenings.

SECONDARY OUTCOMES:
melatonin profile of patients with SOD | 12 months
  For each subject, blood and and saliva samples will be collected and Serum and salivary concentrations of melatonin and of its main metabolite 6-hydroxymelatonin will be measured in samples collected from all patients by using a validated LC-MS method with minor modifications (Magliocco et al 2021).
Sleep EEG description of patients with SOD | 12 months
  A Sleep EEG recording will also be scheduled at the time of study inclusion/evaluation. Previously performed EEG will be revised. EEG assessment will include the analysis of background activity, presence/absence of physiological sleep elements, interictal discharges, sleep macrostructure and microstructure ( spindle characteristics).

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Casimiro Mondino Foundation, Pavia, PV, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pasca L, Morelli F, Catalano G, Quaranta CA, Vitali H, Ballante E, Dattrino F, Crema F, Rota P, Varesio C, De Giorgis V, Romaniello R, Signorini S, Franco V. Sleep profile in patients with septo-optic-pituitary dysplasia: protocol for a prospective cohort study. BMJ Open. 2025 Jan 15;15(1):e090675. doi: 10.1136/bmjopen-2024-090675. PMID 39819934